CLINICAL TRIAL: NCT00287612
Title: Prospective Trial Comparing Utility of Esophageal Crural Dissection During Laparoscopic Fundoplication in Children
Brief Title: Necessity of Esophageal Dissection During Laparoscopic Fundoplication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Shawn St. Peter, Children's Mercy Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05 12-150
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-03

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia
Keywords: GERD; Hiatal Hernia; Recurrence
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Arms:Lap. Fundo. with Mobilization of the Esophageal Junction
  Interventions: Procedure: Lap. Fundo. with Mobilization of the Esophageal Junction
- 2 (Experimental)
  Interventions: Procedure: Lap. Fundo. without Mobilization of the Esophageal Junction

INTERVENTIONS:
Procedure: Lap. Fundo. with Mobilization of the Esophageal Junction — Complete mobilization of the esophageal junction
  Arms: 1
Procedure: Lap. Fundo. without Mobilization of the Esophageal Junction — phrenoesophageal membrane left intact
  Arms: 2

SUMMARY:
This study compares complete dissection of the tissue around the lower esophagus to no dissection of these tissues during laparoscopic fundoplication in children.

DETAILED DESCRIPTION:
This will be a 2-center, prospective randomized clinical trial involving patients who require an operation for gastroesophageal reflux disease. This is intended to be a definitive study. All patients will receive the standard operation for reflux: laparoscopic fundoplication. The dissection will be performed by either separating the phrenoesophageal membrane, or by leaving the phrenoesophageal membrane intact.

Sample size calculated on a power of 80% with an alpha level of 0.05 using the recurrence rates demonstrated by our retrospective data produce a number of 159 patients in each arm of the study. Given that we will need to follow these patients for 1 year after enrollment, there may be some attrition due to lost follow-up. Therefore 180 patients per arm would account for just over 10% attrition.

One group will undergo laparoscopic fundoplication with complete mobilization of the lower esophagus by circumferentially dividing the phrenoesophageal membrane. The other group will undergo laparoscopic fundoplication without dividing this membrane. The operation, post-operative care, and follow-up plan will otherwise not differ between groups.

If 4 consecutive recurrences are found in one group, an interim analysis will be conducted. If a recurrence difference between groups of statistical significance is detected, the study will be concluded at this point. Without this occurrence, an interim analysis will be conducted at 180 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years of age
* Gastroesophageal Reflux Disease

Exclusion Criteria:

1. Hiatal hernia demonstrated on preoperative contrast study, computed tomography or endoscopy
2. Prior esophageal operation (e.g. esophageal atresia repair, esophageal myotomy)
3. Prior operation for congenital diaphragmatic hernia
4. Patient or family circumstance that will create difficulty attaining one-year follow-up (e.g. referral from distance or anticipated relocation of family)
5. Patients not considered laparoscopic candidates by the staff surgeon or anesthesiologist (e.g. carbon dioxide retaining lung disease, congenital heart disease, or complex previous abdominal operations)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2006-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Hiatal hernia | 1 year

SECONDARY OUTCOMES:
control of symptoms | 1 year
retching | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (2):
- United States (2):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Mercy Hospital, Kansas City, Missouri

REFERENCES:
- [Derived] van der Does de Willebois EML; SPICY study group. Mesenteric SParIng versus extensive mesentereCtomY in primary ileocolic resection for ileocaecal Crohn's disease (SPICY): study protocol for randomized controlled trial. BJS Open. 2022 Jan 6;6(1):zrab136. doi: 10.1093/bjsopen/zrab136. PMID 35171266